CLINICAL TRIAL: NCT03341117
Title: Acetylsalicylic Acid Administered in Patients With Type 2 Diabetes Mellitus and Its Effect on the Antioxidant Enzyme System
Brief Title: Acetylsalicylic Acid and Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Sara Pascoe Gonzalez, PhD Clinical Research, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2345
Record Dates: First submitted 2017-09-22; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2; Antioxidant Enzyme System
Keywords: acetylsalicylic acid; antioxidant enzyme system; stress oxidative; type 2 diabetes mellitus.
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: A randomized double blind, placebo controlled clinical trial was carried out in 21 drug naïve adults (35-50 year of age) with DM2 with <5 years since diagnosis. They were overweight or obese (BMI 25.0 - 35.0 kg/m2), had glycosylated hemoglobin A1C (HbA1c) level between 6.5 - 9%. This protocol study was reviewed and approved by the hospital based ethics committee, and written informed consent was obtained from all volunteers. Subject was selected from the same residential area and socioeconomic status. No participants were excessively sedentary or participated in heavy physical activity. All individuals were nonsmokers. Their body weight was stable for al last 3 months before the study.
Who Masked: Participant, Investigator
Masking Description: A randomized double blind, placebo controlled clinical trial was carried out in 21 drug naïve adults,regimen was prescribed to the subjects.
  The allocation was 1:1 concealed and done by simple randomization using a table of random numbers. After randomization, 11 patients received of ASA 300 mg once daily and 10 patients received placebo (calcined magnesia) in the same pharmacological presentation for 90 days, the dose was based in the non-affectation of renal uric acid resorption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylsalicylic acid (Active Comparator): The patients were randomly assigned to received Acetylsalicylic acid 300 mg once daily for 90 days
  Interventions: Drug: Acetylsalicylic acid
- calcined magnesia (Placebo Comparator): The patients were randomly assigned to received placebo (calcinaned magnesia),
  1 capsule 300 mg before each meal for a period of 90 days.
  Interventions: Drug: Calcined magnesia

INTERVENTIONS:
Drug: Acetylsalicylic acid — Acetylsalicylic acid 300 mg per capsule
  Other Names: Aspirin
  Arms: Acetylsalicylic acid
Drug: Calcined magnesia — Calcined magnesia 300 mg per capsule
  Other Names: Placebo
  Arms: calcined magnesia

SUMMARY:
OBJETIVE To assess the effect of acetylsalicylic acid on antioxidant enzymatic system in patients with type 2 diabetes

DETAILED DESCRIPTION:
A randomized, double blind placebo controlled clinical trial was carried out in 21 adult patients with type 2 diabetes. Acetylsalicylic acid 300mg/d was administered orally for 3 months to study group (n=11) and placebo to the control group (n=10).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* BMI 25.0 - 35.0 kg/m2
* HbA1c between 6.5 - 9%.
* Written informed consent
* Same residential area and socioeconomic status.

Exclusion Criteria:

* Sedentary or heavy physical activity.
* Nonsmokers.
* Body weight was stable for al last 3 months before the study.
* Personal history of hepatic, renal, gastric or coronary artery disease.
* Hypersensibility to acetylsalicylic acid.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Modification in the antioxidant enzymatic system activity (total antioxidant capacity, catalase, glutathione peroxidase , superoxide dismutase) in patients with type 2 diabetes after the administration of acetylsalicylic acid | 90 days
  In both groups (intervention an d placebo) of 21 patients each, all the patients with type 2 diabetes mellitus, the antioxidant enzymatic system activity was measured before and after the administration of the acetylsalicylic acid, one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.

SECONDARY OUTCOMES:
Modification in lipid profile in patients with type 2 diabetes after the administration of Acetylsalicylic Acid | 90 days
  In both groups (intervention and placebo ) of 21 patients each , all patients with type 2 diabetes mellitus, lipid profile was measured in mg/dL, before and after the administration of the acetylsalicylic acid, one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.
Hepatic safety after the administration of acetylsalicylic acid through the determination of hepatic profile | 90 days
  The hepatic profile was determined through the serum levels of transaminases in U/L (Glutamic oxalacetic transaminase and Glutamic pyruvic transaminase) after of administration during 90 days of acetylsalicylic acid, The patient was on a 12-hour fast.
Renal safety of administration of acetylsalicylic acid through the determination of serum creatinine | 90 days
  The serum creatinine was measured in mg/dL, before and after of administration during 90 days of acetylsalicylic acid. The patient was on a 12-hour fast.
Modification in HbA1c in patients with type 2 diabetes after the administration of Acetylsalicylic Acid | 90 days
  In both groups (intervention and placebo ) of 21 patients each , all patients with type 2 diabetes mellitus, HbA1c was measured in %, before and after the administration of the acetylsalicylic acid, one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.
Modification in fasting glucose in patients with type 2 diabetes after the administration of Acetylsalicylic acid | 90 days
  In both groups (intervention and placebo ) of 21 patients each , all patients with type 2 diabetes mellitus, glucose was measured in mg/dL, before and after the administration of the acetylsalicylic acid, one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jandeleit-Dahm K, Cooper ME. The role of AGEs in cardiovascular disease. Curr Pharm Des. 2008;14(10):979-86. doi: 10.2174/138161208784139684. PMID 18473849
- [Background] Rahimi R, Nikfar S, Larijani B, Abdollahi M. A review on the role of antioxidants in the management of diabetes and its complications. Biomed Pharmacother. 2005 Aug;59(7):365-73. doi: 10.1016/j.biopha.2005.07.002. PMID 16081237
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Henriksen EJ, Diamond-Stanic MK, Marchionne EM. Oxidative stress and the etiology of insulin resistance and type 2 diabetes. Free Radic Biol Med. 2011 Sep 1;51(5):993-9. doi: 10.1016/j.freeradbiomed.2010.12.005. Epub 2010 Dec 13. PMID 21163347
- [Background] Johansen JS, Harris AK, Rychly DJ, Ergul A. Oxidative stress and the use of antioxidants in diabetes: linking basic science to clinical practice. Cardiovasc Diabetol. 2005 Apr 29;4:5. doi: 10.1186/1475-2840-4-5. PMID 15862133
- [Background] Zatalia SR, Sanusi H. The role of antioxidants in the pathophysiology, complications, and management of diabetes mellitus. Acta Med Indones. 2013 Apr;45(2):141-7. PMID 23770795
- [Background] Newsholme P, Haber EP, Hirabara SM, Rebelato EL, Procopio J, Morgan D, Oliveira-Emilio HC, Carpinelli AR, Curi R. Diabetes associated cell stress and dysfunction: role of mitochondrial and non-mitochondrial ROS production and activity. J Physiol. 2007 Aug 15;583(Pt 1):9-24. doi: 10.1113/jphysiol.2007.135871. Epub 2007 Jun 21. PMID 17584843
- [Background] Lapshina EA, Sudnikovich EJ, Maksimchik JZ, Zabrodskaya SV, Zavodnik LB, Kubyshin VL, Nocun M, Kazmierczak P, Dobaczewski M, Watala C, Zavodnik IB. Antioxidative enzyme and glutathione S-transferase activities in diabetic rats exposed to long-term ASA treatment. Life Sci. 2006 Oct 4;79(19):1804-11. doi: 10.1016/j.lfs.2006.06.008. Epub 2006 Jun 15. PMID 16815474
- [Background] Baltazar MT, Dinis-Oliveira RJ, Duarte JA, Bastos ML, Carvalho F. Antioxidant properties and associated mechanisms of salicylates. Curr Med Chem. 2011;18(21):3252-64. doi: 10.2174/092986711796391552. PMID 21671857
- [Background] Caballero F, Gerez E, Batlle A, Vazquez E. Preventive aspirin treatment of streptozotocin induced diabetes: blockage of oxidative status and revertion of heme enzymes inhibition. Chem Biol Interact. 2000 Jun 1;126(3):215-25. doi: 10.1016/s0009-2797(00)00168-x. PMID 10862819
- [Background] Jeyaseelan L, Rao PS. Methods of determining sample sizes in clinical trials. Indian Pediatr. 1989 Feb;26(2):115-21. PMID 2753525
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Blakytny R, Harding JJ. Prevention of cataract in diabetic rats by aspirin, paracetamol (acetaminophen) and ibuprofen. Exp Eye Res. 1992 Apr;54(4):509-18. doi: 10.1016/0014-4835(92)90129-g. PMID 1623937
- [Background] Coudray C, Favier A. Determination of salicylate hydroxylation products as an in vivo oxidative stress marker. Free Radic Biol Med. 2000 Dec;29(11):1064-70. doi: 10.1016/s0891-5849(00)00403-2. PMID 11121712
- [Background] Ames PR, Batuca JR, Muncy IJ, De La Torre IG, Pascoe-Gonzales S, Guyer K, Matsuura E, Lopez LR. Aspirin insensitive thromboxane generation is associated with oxidative stress in type 2 diabetes mellitus. Thromb Res. 2012 Sep;130(3):350-4. doi: 10.1016/j.thromres.2012.03.025. Epub 2012 Apr 20. PMID 22521214
- [Background] Lemkes BA, Bahler L, Kamphuisen PW, Stroobants AK, Van Den Dool EJ, Hoekstra JB, Nieuwland R, Gerdes VE, Holleman F. The influence of aspirin dose and glycemic control on platelet inhibition in patients with type 2 diabetes mellitus. J Thromb Haemost. 2012 Apr;10(4):639-46. doi: 10.1111/j.1538-7836.2012.04632.x. PMID 22252020
- [Background] Muller KA, Chatterjee M, Rath D, Geisler T. Platelets, inflammation and anti-inflammatory effects of antiplatelet drugs in ACS and CAD. Thromb Haemost. 2015 Aug 31;114(3):498-518. doi: 10.1160/TH14-11-0947. Epub 2015 Jul 30. PMID 26224127
- [Background] Nagelschmitz J, Blunck M, Kraetzschmar J, Ludwig M, Wensing G, Hohlfeld T. Pharmacokinetics and pharmacodynamics of acetylsalicylic acid after intravenous and oral administration to healthy volunteers. Clin Pharmacol. 2014 Mar 19;6:51-9. doi: 10.2147/CPAA.S47895. eCollection 2014. PMID 24672263
- [Background] Dzeshka MS, Shantsila A, Lip GY. Effects of Aspirin on Endothelial Function and Hypertension. Curr Hypertens Rep. 2016 Nov;18(11):83. doi: 10.1007/s11906-016-0688-8. PMID 27787837
- [Background] Grimaldi R, Bisi M, Lonni E, Beggiato E, Valpreda A, Lococo MF, Dosio E, Presutti DG, Tagliabue M, Gaita F. Laboratory aspirin resistance reversibility in diabetic patients: a pilot study using different pharmaceutical formulations. Cardiovasc Drugs Ther. 2014 Aug;28(4):323-9. doi: 10.1007/s10557-014-6536-7. PMID 24984883
- [Background] Abdin AA, Baalash AA, Hamooda HE. Effects of rosiglitazone and aspirin on experimental model of induced type 2 diabetes in rats: focus on insulin resistance and inflammatory markers. J Diabetes Complications. 2010 May-Jun;24(3):168-78. doi: 10.1016/j.jdiacomp.2009.01.005. Epub 2009 Mar 27. PMID 19328014